CLINICAL TRIAL: NCT06247332
Title: Retrospective Data Collection for SENSING-AI: a Wearable Platform for the Early Diagnosis of Emotional Disorders and Exacerbations in Patients With Long COVID Through the Use of Artificial Intelligence
Brief Title: SENSING-AI in Patients With Long COVID (SENSING-AI)
Acronym: SENSING-AI
Status: Completed | Type: Observational
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: SEN-0121
Record Dates: First submitted 2024-01-31; First posted 2024-02-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-02

CONDITIONS: Post-acute COVID-19 Syndrome
Keywords: Long COVID-19; Retrospective study; Artificial Intelligence; Mental Health
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective Long COVID cases: The target population will be as balanced as possible between subjects who needed specialized care due to long COVID-19 complications (either specialized care consultations or any non-planned hospital admission) at 1 month, 3 months, 6 months and 1 year from the long COVID-19 diagnose and those who did not require such specialized care.
  Interventions: Other: Review of available clinical data sources related to use cases

INTERVENTIONS:
Other: Review of available clinical data sources related to use cases — There will be a review of available clinical data sources related to use cases. In addition, this information will be complemented by a cohort of anonymized retrospective data of 100 cases obtained from the clinical information resulting from the assistance to COVID-19 patients managed by the Primary Care Health District of Sevilla Norte and the Infectious Diseases Department of the Virgen Macarena University Hospital

SUMMARY:
The retrospective study will be used to develop an artificial intelligence model of risk stratification of physiological and psychological complications arising from the information available in the electronic medical record and first consultation report to support patients and healthcare professionals in better managing the healthcare process for patients diagnosed with long COVID.

DETAILED DESCRIPTION:
The stratification of the risk of complications related to persistent COVID both physiological and psychological in a personalized way would optimize the cost-effectiveness model for the management of these patients. Similarly, the early detection of complications associated with persistent COVID in patients belonging to vulnerable groups would improve care times and, therefore, the patient's prognosis.

The primary objective for this study is to gather anonymized retrospective data of patients suffering from long COVID in order to contribute to the generation of the SENSING-AI cohort.

ELIGIBILITY:
Inclusion Criteria:

* Legal adult
* Diagnosed of long COVID-19 in the last year
* With the presence of any of these symptoms:
* Asthenia (Tiredness)
* Dyspnea
* Shortness of breath
* Anxiety
* Stress
* Depression
* Sleep disorder

Exclusion Criteria:

* Attended to specialized care consultation
* Was admitted in hospital in the last year due to a problem not related to the COVID complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size for the retrospective study enough to generate a first version of the risk stratification models will be around 100 cases. The target population will be as balanced as possible between subjects who needed specialized care due to long COVID-19 complications (either specialized care consultations or any non-planned hospital admission) at 1 month, 3 months, 6 months and 1 year from the long COVID-19 diagnose and those who did not require such specialized care.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Retrospective SENSING-AI cohort | 1 month
  The retrospective SENSING-AI cohort will be fed from clinical information of 100 cases of patients with long COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Virgen Macarena University Hospital, Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No